CLINICAL TRIAL: NCT01934322
Title: Case Management for Frequent Users of the Emergency Department: A Randomized Controlled Trial
Brief Title: Case Management for Frequent Users of the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Dr Patrick Bodenmann, PD, MER, MSc, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FNS 30023B_135762/1
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Frequent Users of the Emergency Department; Vulnerable Populations
Keywords: frequent users of the emergency department; vulnerable populations; case management; cost savings intervention; quality of life; number of emergency department visits
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case Management (Experimental): Furnish specific assistance and to provide referrals for the patients:
  * If the social determinants are not adequate, the team will lend assistance for obtaining income entitlements, health insurance coverage if eligible, stable housing, schooling for children, etc.
  * If there are mental disturbances, the team will refer to mental health departments inside the hospital, and if necessary, to a psychiatrist, psychologist or general practitioner (GP) out in the community.
  * If the patient presents risk behaviors, the team will refer to substance abuse services and links to community services in order to maintain continuity of care.
  * In case of somatic problems, the team will find a new GP or make contact with the previous provider, contingent on the patient's consent.
  Interventions: Other: Case Management
- Control (No Intervention): Patients randomized to control group (usual care) will receive standard emergency care by physicians (resident or attending physician) and nurses, without the case manager been involved. Nevertheless, the mobile team will take contact with each patient of the control group, giving them short information through a flyer (flyer) which will underline the existence of the mobile team, its addresses and telephone numbers.

INTERVENTIONS:
Other: Case Management — Furnish specific assistance and to provide referrals for the patients:
  * If the social determinants are not adequate, the team will lend assistance for obtaining income entitlements, health insurance coverage if eligible, stable housing, schooling for children, etc.
  * If there are mental disturbances, the team will refer to mental health departments inside the hospital, and if necessary, to a psychiatrist, psychologist or general practitioner (GP) out in the community.
  * If the patient presents risk behaviors, the team will refer to substance abuse services and links to community services in order to maintain continuity of care.
  * In case of somatic problems, the team will find a new GP or make contact with the previous provider, contingent on the patient's consent.
  Arms: Case Management

SUMMARY:
The purpose of this study is to evaluate a specific case management intervention for frequent users (FU) of Emergency Department (ED).

Compared to infrequent or non-users, most of the ED-FU visitors are identified as vulnerable patients because they are more likely to be of low social and economical status, be more isolated and live alone. They report more chronic medical conditions, have a higher mortality rate and consume more healthcare resources.

In the literature, interventions aimed at improving the management of ED-FU have demonstrated several positive outcomes, but there are still some knowledge gaps.

The proposed project tests the hypotheses that case management intervention as compared with standard emergency care

* is a more efficient use of healthcare resources and reduces ED attendance,
* is cost-saving and
* improves quality of life,
* altogether leading to favorable cost-utility ratio.

ELIGIBILITY:
Inclusion Criteria:

* 5 or more attendances during the previous 12 months at the Emergency Department of the University Hospital of Lausanne
* Be capable of communicating in any of the languages spoken by the team (i.e. French, English, German, Italian and Spanish) or through a community interpreter

Exclusion Criteria:

* Patients who cannot give informed consent or are ineligible to receive Case Managers services (e.g. acutely confused, acutely psychotic, intoxicated)
* Patients who are in prison
* Patients with a diagnose of cognitive disorders (delirium, dementia, and other cognitive disorders)
* Patients who are not expected to survive at least 18 months after enrollment
* Patients who will not remain in Switzerland for 12 to 18 months after enrollment
* Family members of a participant already included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
number of Emergency Department visits | 12 months after enrollement

SECONDARY OUTCOMES:
total costs of the healthcare resource | 12 months after enrollement
  costs concerning services provided by the University Hospital of Lausanne and cost concerning services used outside the Hospital

OTHER OUTCOMES:
Quality of life | Day of enrollement, 2 months, 5.5 months, 9 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bodenmann Patrick, PD, MER, MSc, Principal Investigator — University of Lausanne
Locations (1):
- University Hospital of Lausanne, Lausanne, Switzerland

REFERENCES:
- [Background] Althaus F, Paroz S, Hugli O, Ghali WA, Daeppen JB, Peytremann-Bridevaux I, Bodenmann P. Effectiveness of interventions targeting frequent users of emergency departments: a systematic review. Ann Emerg Med. 2011 Jul;58(1):41-52.e42. doi: 10.1016/j.annemergmed.2011.03.007. PMID 21689565
- [Background] Bieler G, Paroz S, Faouzi M, Trueb L, Vaucher P, Althaus F, Daeppen JB, Bodenmann P. Social and medical vulnerability factors of emergency department frequent users in a universal health insurance system. Acad Emerg Med. 2012 Jan;19(1):63-8. doi: 10.1111/j.1553-2712.2011.01246.x. Epub 2012 Jan 5. PMID 22221292
- [Background] Althaus F, Stucki S, Guyot S, Trueb L, Moschetti K, Daeppen JB, Bodenmann P. Characteristics of highly frequent users of a Swiss academic emergency department: a retrospective consecutive case series. Eur J Emerg Med. 2013 Dec;20(6):413-9. doi: 10.1097/MEJ.0b013e32835e078e. PMID 23337095
- [Background] Shumway M, Boccellari A, O'Brien K, Okin RL. Cost-effectiveness of clinical case management for ED frequent users: results of a randomized trial. Am J Emerg Med. 2008 Feb;26(2):155-64. doi: 10.1016/j.ajem.2007.04.021. PMID 18272094
- [Derived] Iglesias K, Baggio S, Moschetti K, Wasserfallen JB, Hugli O, Daeppen JB, Burnand B, Bodenmann P. Using case management in a universal health coverage system to improve quality of life of frequent Emergency Department users: a randomized controlled trial. Qual Life Res. 2018 Feb;27(2):503-513. doi: 10.1007/s11136-017-1739-6. Epub 2017 Nov 29. PMID 29188481
- [Derived] Bodenmann P, Velonaki VS, Ruggeri O, Hugli O, Burnand B, Wasserfallen JB, Moschetti K, Iglesias K, Baggio S, Daeppen JB. Case management for frequent users of the emergency department: study protocol of a randomised controlled trial. BMC Health Serv Res. 2014 Jun 17;14:264. doi: 10.1186/1472-6963-14-264. PMID 24938769